CLINICAL TRIAL: NCT07130019
Title: Autofluorescence-Guided Removal of Psoriatic Tissue
Brief Title: Is Monitoring Enhanced Auto-fluorescence Beneficial for the Precise Removal of Tissue From Psoriatic Lesions With Ablative Lasers?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nick van der Beek (Other)
Responsible Party: Sponsor-Investigator, Nick van der Beek, General manager, ZBC MultiCare
Organization: ZBC MultiCare (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPA-2
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: psoriasis; lasertherapy; fluorescence
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluorescence controlled ablation (Experimental): Fluorescence guided thermal tissue ablation
  Interventions: Procedure: Fluorescence guided thermal ablation of epidermal tissue
- Classic tissue ablation (Active Comparator): Thermal tissue ablation a vue
  Interventions: Procedure: Thermal ablation of epidermal tissue
- Control (No Intervention)

INTERVENTIONS:
Procedure: Fluorescence guided thermal ablation of epidermal tissue — Thermal ablation of epidermal tissue under fluorescence control.
  Arms: Fluorescence controlled ablation
Procedure: Thermal ablation of epidermal tissue — Thermal ablation of skin tissue a vue
  Arms: Classic tissue ablation

SUMMARY:
It is known that psoriatic lesions clear and remain cleared if you remove them from the skin. This can be done through surgery and ablative laser therapy. In order for the treatment to be succesful, you need to remove the complete epidermis and a bit of the dermis (the upper part of the skin). In psoriasis, the thickness of that part of the skin can vary significantly. Incomplete removal results in the return of the lesion. A challenge is that you can't easily tell how deep into the skin you are. Not only is the skin quite thin (from 0.1 mm to 1.0 mm), at the boundary they look quite similar. If you go too deep, you get scarring. Thus there is a need to delineate the psoriatic tissue from the healthy tissue.

We think that one way to do that is by looking at the fluorescence of the skin. If you shine a particular shade of blue light on the skin, it gives off red light. But this is only true for the part where the psoriasis can reside. Under normal circumstances this fluorescence is too weak to really see with the eye. Thus we first increase the fluorescence by administering a compound that is used to make the fluorescent molecules in our tissue, 5-aminolevulinic acid (5-ALA). It can be quite difficult to get 5-ALA into the skin. To help the 5-ALA, we use a very superficial lasertreatment to poke minute holes in the skin. The 5-ALA enters the skin and the fluorescence builds up. After a couple of hours, the skin is treated with a laser that can gently remove the tissue. Layer for layer is removed until there is no more fluorescence. At that point we do one more pass to be sure, and then stop. We hope that two months later, the psoriasis is gone and will remain so for at least a year.

We think that the fluorescence helps, but we can't be sure. So for that reason we will also treat a lesion without fluorescence and use the standard method to judge how deep we have treated the skin. And to rule out the possibility that e.g. sun exposure cleared the lesions, we also leave one lesion untreated.

Participants have to travel to the clinic for the treatment and then every three to five days for two weeks. Since we remove the skin, there will be a wound that needs healing and attending to. This will result in some limitations during the wound healing phase. Afterwards, you might see some temporary shifts in pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psoriasis vulgaris of any severity with at least three discrete lesions in optically non-obscured skin located on torso, abdomen, dorsum, legs, arms, face or buttocks.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Rheumatoid and psoriatic arthritis
* Fitzpatrick skin type >4.
* Known allergy to 5-aminolevulinic acid (5-ALA) or light sensitivity.
* Autoimmune disorders.
* Heavy smoking.
* Diabetes mellitus type 2
* Active bacterial or viral infections in the treatment area
* Recent use of isotretinoin
* Morbid obesity
* History of hypertrophic scaring or keloids
* History of complicated wound healing
* Body dysmorphic disorder
* Use of anti-coagulants
* Use of cyclosporin A or similar immunosuppressive medication
* Increase in disease severity during the preceding 8 weeks.
* If treatment area is on the legs: Severe venous insufficiency, severe lymphoedema or angiopathy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
PGA | 8 weeks
  PGA value (0 - 7)
Remission | 8 weeks
  Remission score (0,1)

SECONDARY OUTCOMES:
Healing time | 8 weeks
  Healing time in weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ZBC Multicare, Hilversum, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
PGA Remission
Supporting Information: Study Protocol, ICF
Access Criteria: Researchers at academic institutions who have a public track record in the field of laser therapy for psoriasis or those who can provide similar qualifications.
  Interested researchers can contact the prinicipal investigator, details provided in this registration.